CLINICAL TRIAL: NCT07074431
Title: "Comparative Study of High-frequency Pulsed Vacuum Technology Versus Phacoemulsification for Cataract Surgery
Acronym: PULSEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Victor Pauchet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-A02793-44
Record Dates: First submitted 2025-05-15; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cataract Bilateral
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECHNIC BY CATAPULSE (Experimental)
  Interventions: Procedure: EYE 1 SURGERY BY CATAPULSE TECHNIC
- TECHNIC BY PHACOEMULSIFICATION (Active Comparator)
  Interventions: Procedure: EYE 2 SURGERY BY CATAPULSE TECHNIC

INTERVENTIONS:
Procedure: EYE 1 SURGERY BY CATAPULSE TECHNIC — In arm 2: 1st eye operated by high-frequency pulsed vacuum technology / 2nd eye operated by phacoemulsification
  Arms: TECHNIC BY CATAPULSE
Procedure: EYE 2 SURGERY BY CATAPULSE TECHNIC — In arm 1: 1st eye operated by phacoemulsification / 2nd eye operated by high-frequency pulsed vacuum technology
  Arms: TECHNIC BY PHACOEMULSIFICATION

SUMMARY:
Cataracts are cloudings of the lens, primarily due to aging. Surgery is the primary treatment for cataracts. The most commonly used surgical technique is phacoemulsification, which involves fragmenting the lens using a high-frequency ultrasound probe and removing the fragments. Phacoemulsification is more common due to its advantages.

Recently, a new approach has emerged, using high-frequency pulsed vacuum technology for cataract ablation. This less invasive approach is expected to allow for faster patient recovery and reduce surgical risks. High-frequency pulsed vacuum utilizes the pulse-pulse principle by interrupting the vacuum every tenth of a second. This interruption creates an impact moment between the cataract material and the cannula tip, dissecting the cataract without damaging the surrounding delicate tissue. High-frequency pulsed vacuum maintains anterior chamber stability while creating sufficient dissection to aspirate the cataract material. This energy also cools the tip, allows for better vacuum control, and significantly reduces turbulence within the eye. More importantly, high-frequency pulsed vacuum disrupts endothelial cells less and causes less edema than mechanical ultrasound.

This technique therefore appears ideal for treating patients with at-risk corneas (low endothelial cell count, risk of decompensation and corneal transplantation).

The objective of the study is to demonstrate the benefits of this approach using high-frequency pulsed vacuum technology through a randomized, comparative, crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient with bilateral cataracts
* Grade 1 to 3 cataracts
* Indication for bilateral cataract surgery
* Patient informed of the study and having given their written and signed informed consent
* Patient affiliated with a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Refusal of consent
* Cataract grade > 3
* Unilateral and/or combined cataract surgery
* Uveitic cataract
* Glaucoma
* Patient with ocular comorbidity
* Patient with cognitive impairment preventing them from responding to satisfaction questionnaires
* Patient unable to read, write, or understand French
* Pregnant or breastfeeding patient as defined in Article L1121-5 of the French Public Health Code
* Vulnerable patient as defined in Article L1121-6 of the French Public Health Code
* Adult patient under guardianship, curatorship, or legal protection
* Patient unable to give personal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell count by specular microscopy after each surgery | At Day30 (+/- 7 days)
  The patient is placed in front of a mirror microscope, the chin resting on a chin rest, the ophthalmologist observes the endothelial layer of the cornea through the microscope, he manually counts the endothelial cells and assesses their density

SECONDARY OUTCOMES:
Visual acuity | before each procedure, between day 1 and day 5 after each procedure, and day 30 (+/- 7 days) after each procedure
  Vision is tested in distance and near vision, eye by eye, by masking with a patch
Measurement of postoperative inflammation | Between Day 1 and Day 5 after each cataract surgery
  The measurement of inflammation is carried out using the SUN classification
The rate of postoperative complications | Between Day 1 and Day 5 after each cataract surgery, at Day30 (+/- 7 days)
The operating times of each surgery | Perioperative
Satisfaction with the use of high-frequency pulsed vacuum technology by healthcare teams | Between Day 1 and Day 5 after each cataract surgery with CATAPULSE
  The satisfaction will be assessed using a questionnaire
A Likert scale will be used to assess patient comfort during surgery | Between Day 1 and Day 5 after each cataract surgery
  The comfort will be assessed using a questionnaire
Adverse events related to both surgeries | Between Day 1 and Day 5 after each cataract surgery and at Day30 (+/- 7 days)

IPD SHARING:
Plan to Share IPD: Undecided